CLINICAL TRIAL: NCT03774407
Title: Dual Benefits of Vaginal Estriol: Improved Urogenital Health and Re-myelination in Relapsing Remitting Multiple Sclerosis (RRMS)
Brief Title: Vaginal Estriol in Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L19-020
Record Dates: First submitted 2018-12-05; First posted 2018-12-13 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis; Neurogenic Bladder
Keywords: remyelination; urogenital health; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: This is a single-group prospective repeated-measures pilot trial. Duration is 12 months,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- urogenital symptoms (Other): To evaluate the efficiency of vaginal estriol, as a treatment for urogenital symptoms in female patients with RRMS.
  Interventions: Drug: vaginal estriol
- remyelination (Experimental): To evaluate the potential role of vaginal estriol in re-myelination in RRMS patients.
  Interventions: Drug: vaginal estriol

INTERVENTIONS:
Drug: vaginal estriol — Estriol vaginal cream will be formulated by Twin Oaks specialty pharmacy-by the same compound specialist. 30 mg estriol powder will be mixed with 5 mL of propylene glycol and 22 g of vaginal base cream. The product can be stored at room temperature and has a shelf life of up to 4 months. It comes with an applicator.
  Other Names: estriol cream

SUMMARY:
Study to evaluate the efficiency of vaginal estriol, as a treatment for urogenital symptoms in female patients with RRMS. The secondary objective is to evaluate the potential role of vaginal estriol in re-myelination in RRMS patients.

DETAILED DESCRIPTION:
Pilot project to determine the effectiveness of 1 mg transvaginal estriol, as an adjunctive therapy for female MS patients. The goal is to recruit 20 patients from the MS clinic in the neurology department of Texas Tech University Health Sciences Center. This study has been planned in collaboration with reproductive endocrinology, endocrinology, gynecology and basic science. The 1mg transvaginal dose was chosen after careful search of the literature and consultation with collaborators.

Single-group pilot study.

Subjects:

Patients with relapsing remitting MS and urogenital symptoms (frequency, urgency, frequent urinary tract infections, incontinence) will be invited to participate in the study. Enrollment will be during their scheduled clinic appointment. Some candidates (patients of the primary investigator) may be contacted by phone and invited to participate in the study.

The clinical trial will be explained to potential participants in detail, reviewing the objectives and methodology of the study. There will be adequate time allotted to answer any questions or concerns from the potential participants. Those patients interested in participating in the study will be asked to sign the consent form. In order to remind patients about their follow-up visits, lab work, etc., they will be contacted routinely. Participants will be instructed to call in case of questions or concerns.

Patients will be evaluated clinically during their scheduled follow up in which a full neurological exam will be performed during each visit. Patients will be instructed by the primary investigator how to correctly use the vaginal cream. This will be done at their enrolment and reinforced by the principal investigator, during their follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with RRMS over the age of 40 to 65.

   * Being prescribed vaginal estriol to treat their urogenital symptoms such as frequency, urgency, incontinence and frequent urinary tract infections.
   * Patients that had underwent chemical or surgical hysterectomy.
2. Patients will continue their current disease modifying agent for MS during the trial.

Exclusion Criteria:

1. Patients with history of breast cancer, uterine or ovarian cancer.
2. Patients with progressive multiple sclerosis
3. Patients who are unable to undergo an MRI
4. Males
5. Patient is already on vaginal or oral or transdermal estrogens
6. Pregnant or breast-feeding patients
7. Patient taking sex hormones eg testosterone for libido
8. Patients taking DHEA or OTC related products that could influence the hormonal milieu.
9. Patient with prolapse uterus or conditions that would impact on transvaginal absorption of estriol

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 21 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirla Avila, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Avila-Ornelas J, Avila M, Stosic M, Robles L, Prieto PG, Hutton GJ, Rivera VM. The role of postpartum intravenous corticosteroids in the prevention of relapses in multiple sclerosis. Int J MS Care. 2011 Summer;13(2):91-3. doi: 10.7224/1537-2073-13.2.91. PMID 24453710
- [Result] Cody JD, Jacobs ML, Richardson K, Moehrer B, Hextall A. Oestrogen therapy for urinary incontinence in post-menopausal women. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD001405. doi: 10.1002/14651858.CD001405.pub3. PMID 23076892
- [Result] Harlow DE, Honce JM, Miravalle AA. Remyelination Therapy in Multiple Sclerosis. Front Neurol. 2015 Dec 10;6:257. doi: 10.3389/fneur.2015.00257. eCollection 2015. PMID 26696956
- [Result] Mallik S, Samson RS, Wheeler-Kingshott CA, Miller DH. Imaging outcomes for trials of remyelination in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2014 Dec;85(12):1396-404. doi: 10.1136/jnnp-2014-307650. Epub 2014 Apr 25. PMID 24769473
- [Result] Moore KH. The costs of urinary incontinence. Med J Aust. 2001 May 7;174(9):436-7. doi: 10.5694/j.1326-5377.2001.tb143368.x. No abstract available. PMID 11386586
- [Result] Rahn DD, Carberry C, Sanses TV, Mamik MM, Ward RM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen for genitourinary syndrome of menopause: a systematic review. Obstet Gynecol. 2014 Dec;124(6):1147-1156. doi: 10.1097/AOG.0000000000000526. PMID 25415166
- [Result] Tiwari-Woodruff S, Voskuhl RR. Neuroprotective and anti-inflammatory effects of estrogen receptor ligand treatment in mice. J Neurol Sci. 2009 Nov 15;286(1-2):81-5. doi: 10.1016/j.jns.2009.04.023. Epub 2009 May 13. PMID 19442988

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: one participant was enrolled twice
Groups:
- Vaginal Estriol as a Potential Adjunctive Therapy for MS Remyelination: Pilot study at TTUHSC department of neurology, MS clinic. Adjunctive vaginal estriol (1mg) was offered to patient with RRMS. MRI brain with and without contrast, VEP and OCT obtained at baseline and 9 months. Multiple sclerosis quality of life-54(MSQOL-54) mental and physical were performed at first encounter and 9 months. Vaginal estriol is absorbed more naturally, levels of FSH, estriol and LH were done at baseline and 9 months. Total 12 patients included.
Period: Overall Study
Arm/Group | Vaginal Estriol as a Potential Adjunctive Therapy for MS Remyelination
Started | 21
Completed | 12
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Vaginal Estriol as a Potential Adjunctive Therapy for MS Remyelination: To evaluate the efficiency of vaginal estriol, as a treatment for urogenital symptoms in female patients with RRMS.
  vaginal estriol: Estriol vaginal cream will be formulated by Twin Oaks specialty pharmacy-by the same compound specialist. 30 mg estriol powder will be mixed with 5 mL of propylene glycol and 22 g of vaginal base cream. The product can be stored at room temperature and has a shelf life of up to 4 months. It comes with an applicator.
Arm/Group | Vaginal Estriol as a Potential Adjunctive Therapy for MS Remyelination
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Bladder Control Scale (BLCS)
Description: The questions are regarding control of the bladder, number of accidents in the past 4 weeks, alteration of activities because of bladder problems and restriction on lifestyle because of bladder problems. The total score for the BLCS is the sum of the scores for the 4 items. Scores can range from 0-22, with higher scores indicating greater bladder control problems. Change from baseline at 9 months.
Time Frame: baseline and 9 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Urogenital Symptoms: Evaluate the efficiency of vaginal estriol, as a treatment for urogenital symptoms in female patients with RRMS.
  vaginal estriol: Estriol vaginal cream will be formulated by Twin Oaks specialty pharmacy-by the same compound specialist. 30 mg estriol powder will be mixed with 5 mL of propylene glycol and 22 g of vaginal base cream. The product can be stored at room temperature and has a shelf life of up to 4 months. It comes with an applicator.
Arm/Group | Urogenital Symptoms
Number analyzed (Participants) | 12
score on a scale | -9 [-11 to -7]
Statistical Analysis 1: Comparison: Urogenital Symptoms; Test type: Other; p = 0.002, p value — This P value reported was for bladder urinary frequency change from baseline to 9 months

2. Primary Outcome: Change in Visual Evoked Potential and Ocular Tomography Results From Baseline to 9 Months of Both Eyes
Description: visual evoked potential measured in each eye at baseline and 9 months normal value should be bellow 100 milliseconds
Time Frame: Baseline and 9 months
Population: patients were evaluated at baseline and 9 months
Measure: Mean (Standard Deviation); unit: millisecond
Groups:
- Ocular Tomography: ocular tomography (evaluates the thickness of the retina) measured in each eye at baseline and 9 months
Arm/Group | Ocular Tomography
Number analyzed (Participants) | 12
millisecond
  R EYE | -4.4 (10.4)
  L EYE | -10.7 (14.4)

3. Primary Outcome: Change in MS Quality of Life Questionnaire at Baseline and 9 Months. (Physical Score)
Description: Multiple sclerosis quality of life questionnaire is an extensive questionnaire filled by the patient and graded by physician. It consists of 2 main areas the physical health which include physical function, health perceptions, energy fatigue, role limitations, pain, sexual function, social function and health distress. The mental health score which includes health distress, overall quality of life, emotional wellbeing, role limitations and cognitive function. The physical health and mental health parts each include a possible score range of 0-100. Overall the lower the score the better
Time Frame: Quality of life score at baseline and Quality of life score at 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Quality of Life Questionnaire: quality of life questionnaire to be compared at baseline and 9 months
Arm/Group | Quality of Life Questionnaire
Number analyzed (Participants) | 12
score on a scale
  Quality of life Physical score | 14.87 (16.9)
  Quality of life Mental score | 10.8 (17.8)

ADVERSE EVENTS:
Time Frame: baseline and 9 months
Description: Between baseline and 9 months
Groups:
- Vaginal Estriol as a Potential Adjunctive Therapy for MS Remyelination: no adverse events were reported
Arm/Group | Vaginal Estriol as a Potential Adjunctive Therapy for MS Remyelination
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03774407/Prot_SAP_002.pdf
  • Informed Consent Form (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03774407/ICF_000.pdf